CLINICAL TRIAL: NCT00559195
Title: Phase 2 Study Evaluating the Efficacy of Epoetin Beta (Neocormon®) For Fatigue and Quality of Life of Patients Receiving Palliative Care for a Solid Malignant Tumor
Brief Title: Epoetin Beta in Treating Fatigue and Anemia in Patients Receiving Palliative Care for Malignant Solid Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Hospital Regional Universitaire de Limoges (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Non-Randomized | Purpose: Supportive Care
Other Study IDs: CDR0000574173; CHUL-NEOPALIA; RECF0359
Record Dates: First submitted 2007-11-15; First posted 2007-11-16 (Estimated); Last update posted 2011-05-16 (Estimated); Status verified 2011-05

CONDITIONS: Anemia; Fatigue; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific; anemia; fatigue
MeSH Terms: conditions — Anemia; Fatigue | interventions — epoetin beta

INTERVENTIONS:
Biological: epoetin beta
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: Epoetin beta may cause the body to make more red blood cells and may help relieve fatigue in patients with malignant solid tumors receiving palliative care.

PURPOSE: This phase II trial is studying how well epoetin beta works in treating fatigue and anemia in patients receiving palliative care for malignant solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Evaluate the impact of epoetin beta on fatigue and quality of life of patients receiving palliative care for malignant solid tumors.

Secondary

* Evaluate the impact of epoetin beta on hemoglobin level (increase > 2 g/dL).

OUTLINE: Patients receive epoetin beta subcutaneously once a week for up to 3 months.

Fatigue, quality of life, and hemoglobin and reticulocyte levels are assessed every 4 weeks.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed malignant solid tumor

  * No hematologic malignancy
* Hemoglobin < 10.5 g/dL (anemic)
* Receiving palliative care only

PATIENT CHARACTERISTICS:

* Life expectancy > 6 months
* Negative pregnancy test
* Fertile patients must use effective contraception
* No chronic anemia requiring treatment (e.g., thalassemia or sickle cell disease)
* No uncontrolled hypertension
* No allergy to any drugs or components used in the study
* Not a prisoner or under guardianship or trusteeship
* No mental disability that impairs a clear understanding of the study requirements

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* More than 2 months since prior specific anticancer therapy (e.g., chemotherapy, hormonal therapy, targeted therapy, or immunotherapy)
* More than 1 month since prior and no concurrent participation in another clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2005-11; Primary Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Fatigue
Quality of life

SECONDARY OUTCOMES:
Hemoglobin level

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Luc Labourey, Study Chair — Centre Hospital Regional Universitaire de Limoges
Locations (1):
- Centre Hospital Regional Universitaire de Limoges, Limoges, France